CLINICAL TRIAL: NCT00481078
Title: Randomized Phase II Study of Vorinostat or Placebo in Combination With Carboplatin and Paclitaxel for Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Vorinostat, Carboplatin, and Paclitaxel in Treating Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02841; PHII-82; N01CM62208 (NIH); N01CM62209 (NIH); N01CM62201 (NIH)
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Paclitaxel; Taxes; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (vorinostat, paclitaxel, carboplatin) (Experimental): Patients receive oral vorinostat (SAHA) at 400 mg once daily on days 1-14 and paclitaxel IV 200 mg/m2 over 3 hours and carboplatin IV dosed to achieve an area under the concentration versus time curve of 6 mg/mLXmin over 30 minutes on day 3.
  Interventions: Drug: vorinostat; Drug: paclitaxel; Drug: carboplatin; Other: laboratory biomarker analysis
- Arm II (placebo, paclitaxel, carboplatin) (Active Comparator): Patients receive an oral placebo once daily on days 1-14 and paclitaxel and carboplatin as in arm l.
  Interventions: Drug: paclitaxel; Drug: carboplatin; Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
  Arms: Arm I (vorinostat, paclitaxel, carboplatin)
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo, paclitaxel, carboplatin)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying carboplatin, paclitaxel, and vorinostat to see how well they work compared with carboplatin, paclitaxel, and a placebo in treating patients with stage III or stage IV non-small cell lung cancer. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving carboplatin and paclitaxel together with vorinostat is more effective than giving carboplatin and paclitaxel together with a placebo in treating non-small cell lung cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the response rate associated with the combination of vorinostat, carboplatin, paclitaxel versus carboplatin, paclitaxel and placebo for patients with previously untreated, advanced NSCLC.

SECONDARY OBJECTIVES:

I. To determine the time to progression and overall survival for the two regimens.

II. To assess the safety profile of the regimen of vorinostat, carboplatin and paclitaxel for patients with advanced NSCLC.

III. To understand mechanistic aspects of drug effect by conducting correlative science studies on peripheral blood, archived tumor tissue, and paired biopsies in consenting patients.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to gender and brain metastasis (present vs absent). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral vorinostat (SAHA) once daily on days 1-14 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 3.

Arm II: Patients receive an oral placebo once daily on days 1-14 and paclitaxel and carboplatin as in arm l.

In both arms, treatment repeats every 21 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed stage IIIB (with malignant pleural pericardial effusion) or stage IV non-small cell lung cancer
* No prior chemotherapy for advanced or metastatic disease
* ECOG performance status 0 or 1
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Vorinostat can cause fetal harm when administered to a pregnant woman; there are no adequate and well-controlled studies in pregnant women; if this drug is used during pregnancy, or if the patient becomes pregnant while taking this drug, the patient should be apprised of the potential hazard to the fetus
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with untreated brain metastases should be excluded from this clinical trial; however, patients who have stable brain disease (should be off corticosteroids) at least 3 weeks after completion of appropriate therapy are eligible
* Prior or current use of valproic acid, a HDAC inhibitor
* Peripheral neuropathy of severity greater than grade 1
* Known history of allergic reactions to paclitaxel
* Prior therapy with paclitaxel
* Inability to take oral medications on a continuous basis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because vorinostat is an HDAC inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, breastfeeding should be discontinued if the mother is treated with vorinostat; these potential risks may also apply to other agents used in this study
* HIV-positive patients receiving combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with vorinostat; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Belani, Principal Investigator — Penn State Hershey Cancer Institute
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Vorinostat, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin)
Started | 62 | 32
Completed | 20 | 12
Not Completed | 42 | 20
Not completed — Progression of disease | 11 | 11
Not completed — Adverse Event | 15 | 3
Not completed — Death | 5 | 3
Not completed — Intercurrent illness | 1 | 0
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Information not available | 1 | 0
Not completed — Received other treatment | 2 | 1
Not completed — Brain metastasis | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Patients receive oral vorinostat (SAHA) at 400 mg once daily on days 1-14 and paclitaxel IV 200 mg/m2 over 3 hours and carboplatin IV dosed to achieve an area under the concentration versus time curve of 6 mg/mLXmin over 30 minutes on day 3.
- Arm 2: Patients receive an oral placebo once daily on days 1-14 and paclitaxel and carboplatin as in arm l.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 62 | 32 | 94
Age, Continuous [Median (Full Range); unit: years] | 64 [32 to 83] | 66.5 [48 to 85] | 65 [32 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 12 | 36
  Male | 38 | 20 | 58
Region of Enrollment [Number; unit: participants]
  United States | 62 | 32 | 94

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Each patient will be assigned one of the following categories: 1) complete response, 2) partial response, 3) stable disease, 4) progressive disease, 5) early death from malignant disease, 6) early death from toxicity, 7) early death because of other cause, or 9) unknown (not assessable, insufficient data).
  Patients with confirmed CR or PR according to the RECIST criteria were considered to have responded to treatment.
Time Frame: Assessed every two cycles
Measure: Number (95% Confidence Interval); unit: percentage of responding patients
Arm/Group | Arm I (Vorinostat, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 62 | 32
percentage of responding patients | 34 [22 to 47] | 12.5 [4 to 29]

2. Secondary Outcome: Progression-free Survival
Description: Evaluated using the Kaplan-Meier method. Compared between arms using the log-rank test.
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Vorinostat, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 62 | 32
Months | 6 [4.3 to 6.9] | 4.1 [1.9 to 5.5]

3. Secondary Outcome: Overall Survival
Description: Evaluated using the Kaplan-Meier method. Compared between arms using the log-rank test.
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Vorinostat, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 62 | 32
Months | 13 [9.7 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 9.7 [6 to 13]

ADVERSE EVENTS:
Description: "Other" adverse events include all grades and attributions to treatment not included in the "Serious" adverse events table.
Arm/Group | Arm I (Vorinostat, Paclitaxel, Carboplatin) | Arm II (Placebo, Paclitaxel, Carboplatin)
Serious Adverse Events (participants affected / at risk) | 29/61 | 10/32
Other Adverse Events (participants affected / at risk) | 61/61 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Vorinostat, Paclitaxel, Carboplatin) (N=61) | Arm II (Placebo, Paclitaxel, Carboplatin) (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 1 (1)
Disease progression (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (5) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 4 (5) | 2 (3)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (6) | 2 (2)
Platelet count decreased (Investigations) | 7 (9) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Personality change (Psychiatric disorders) | 1 (1) | 1 (2)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 2 (3)
Thrombosis (Vascular disorders) | 2 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Vorinostat, Paclitaxel, Carboplatin) (N=61) | Arm II (Placebo, Paclitaxel, Carboplatin) (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 43 (126) | 21 (71)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (3) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (5) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (7) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (3) | 2 (2)
Watering eyes (Eye disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (11) | 2 (3)
Constipation (Gastrointestinal disorders) | 23 (43) | 13 (26)
Diarrhea (Gastrointestinal disorders) | 20 (39) | 8 (20)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 5 (7) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 4 (7) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 7 (9) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (6) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (3) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 2 (4) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 37 (77) | 14 (30)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 25 (36) | 5 (10)
Chest pain (General disorders) | 9 (15) | 2 (2)
Chills (General disorders) | 7 (8) | 1 (2)
Death (General disorders) | 5 (5) | 6 (6)
Disease progression (General disorders) | 20 (20) | 14 (14)
Edema limbs (General disorders) | 7 (19) | 5 (10)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 52 (115) | 21 (61)
Fever (General disorders) | 8 (8) | 4 (5)
Gait abnormal (General disorders) | 1 (1) | 0 (0)
General symptom (General disorders) | 1 (1) | 1 (2)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 3 (4)
Localized edema (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 4 (4) | 2 (3)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Bladder infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (3) | 1 (1)
Mucosal infection (Infections and infestations) | 2 (2) | 0 (0)
Opportunistic infection (Infections and infestations) | 1 (1) | 0 (0)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (15) | 4 (7)
Alkaline phosphatase increased (Investigations) | 13 (28) | 7 (20)
Aspartate aminotransferase increased (Investigations) | 9 (19) | 3 (4)
Bilirubin increased (Investigations) | 5 (10) | 1 (4)
Creatine phosphokinase increased (Investigations) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 7 (21) | 1 (2)
INR increased (Investigations) | 2 (4) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 28 (66) | 14 (31)
Lymphocyte count decreased (Investigations) | 14 (43) | 7 (14)
Neutrophil count decreased (Investigations) | 31 (60) | 17 (36)
Platelet count decreased (Investigations) | 36 (87) | 15 (38)
Serum cholesterol increased (Investigations) | 1 (4) | 0 (0)
Weight loss (Investigations) | 10 (16) | 4 (13)
Anorexia (Metabolism and nutrition disorders) | 35 (57) | 11 (24)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 5 (9) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 29 (79) | 15 (39)
Dehydration (Metabolism and nutrition disorders) | 10 (15) | 3 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 18 (36) | 6 (21)
Serum calcium decreased (Metabolism and nutrition disorders) | 17 (28) | 3 (6)
Serum calcium increased (Metabolism and nutrition disorders) | 5 (7) | 2 (5)
Serum glucose decreased (Metabolism and nutrition disorders) | 4 (7) | 2 (4)
Serum magnesium decreased (Metabolism and nutrition disorders) | 6 (15) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 10 (21) | 3 (4)
Serum potassium decreased (Metabolism and nutrition disorders) | 13 (21) | 7 (17)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 18 (36) | 9 (14)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 3 (8)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (17) | 1 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5)
Joint pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 6 (13)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (12) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (20) | 6 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (21) | 2 (4)
Arachnoiditis (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 3 (4) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 16 (23) | 6 (7)
Headache (Nervous system disorders) | 6 (9) | 4 (6)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 29 (87) | 12 (33)
Phantom pain (Nervous system disorders) | 0 (0) | 1 (3)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Taste alteration (Nervous system disorders) | 11 (23) | 4 (5)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 1 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (6) | 3 (4)
Confusion (Psychiatric disorders) | 6 (11) | 3 (4)
Depression (Psychiatric disorders) | 3 (5) | 3 (5)
Insomnia (Psychiatric disorders) | 10 (17) | 5 (11)
Personality change (Psychiatric disorders) | 2 (2) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (3) | 1 (3)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (3) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 2 (7) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (3) | 1 (2)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (15) | 2 (7)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (40) | 9 (23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (34) | 7 (15)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (1)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (57) | 10 (32)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (8) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 7 (11) | 7 (10)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 6 (10) | 3 (5)
Phlebitis (Vascular disorders) | 1 (1) | 1 (2)
Thrombosis (Vascular disorders) | 1 (3) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less